CLINICAL TRIAL: NCT03284788
Title: Wellness Achieved Through Changing Habits (The WATCH Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: StayWell (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); WellCare Health Plans, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701609-N; K01HL141535 (NIH); PA-16-190 (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2017-08-29; First posted 2017-09-15 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Weight Loss; Obesity; Overweight
Keywords: acceptance-based therapy; adolescents; weight; weight loss; obesity; overweight
MeSH Terms: conditions — Weight Loss; Obesity; Overweight; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABT Weight Loss Intervention (Experimental): Adolescent girls will attend healthy lifestyle sessions that include nutritional education and physical activity education and build skills in the areas of values clarification, mindfulness, self-regulation skills, acceptance of uncomfortable states, goal-setting, problem solving, and self-monitoring.
  Interventions: Behavioral: ABT Weight Loss Intervention

INTERVENTIONS:
Behavioral: ABT Weight Loss Intervention — This includes 15 sessions that are each 90 minutes in length. Intervention sessions will be weekly for the first 2 months, bi-weekly for the next 2 months, and monthly for the last 2 months.

SUMMARY:
The purpose of this pilot, feasibility study is to investigate the acceptability of an acceptance-based therapy healthy lifestyle intervention in adolescent girls with overweight/obesity.

DETAILED DESCRIPTION:
Participants will attend 2 baseline clinic visits and adolescents will participate in an ABT healthy lifestyle intervention.

The intervention will include 15 sessions over 6 months.

A post-treatment visit will occur.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls between ages 14-19 with overweight or obesity above the 85th percentile for sex and age as determined by CDC growth charts

Exclusion Criteria:

* Known pregnancy or plans to become pregnant in the next 2 years
* Any condition prohibiting physical activity
* A diagnosis of cardiovascular disease or diabetes
* Have active cancer or cancer requiring treatment in the past 2 years
* Have active or chronic infections (e.g., HIV or TB)
* Have active kidney disease or lung disease
* An eating disorder or substance abuse disorder
* Having begun a course of or changed the dosage of any medications known to affect appetite or body composition within the previous 3 months
* Weight loss greater than or equal to 5% in the previous 6 months
* If they do not follow the study plan

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle I Cardel, PhD, MS, RD, Principal Investigator — University of Florida
Locations (1):
- HealthStreet and University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in clinics or through social media.
Pre-assignment Details: 60 participants were screened for eligibility. Of these 43 were excluded (n=12 did not meet inclusion criteria, 31 declined to participate). 17 participants consented; 16 completed the baseline visits. 13 decided to participate in the intervention.
Groups:
- ABT Intervention: Participants attended 15, 90-minute sessions via videoconferencing software. They also met with a registered dietitian at baseline.
Period: Overall Study
Arm/Group | ABT Intervention
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- ABT Intervention: Adolescent girls will attend healthy lifestyle sessions that include nutritional education and physical activity education and build skills in the areas of values clarification, mindfulness, self-regulation skills, acceptance of uncomfortable states, goal-setting, problem solving, and self-monitoring.
Arm/Group | ABT Intervention
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.69 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 2
  Not Hispanic/Latina | 11
  White | 7
  Black | 5
  Multiple Races | 1
Highest parental education [Count of Participants; unit: Participants]
  High school diploma/GED | 2
  Some college/associate degree | 3
  College graduate | 3
  Graduate or professional degree | 4
  Unknown | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.28 (5.50)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: Number of teens who enrolled and completed both initial baseline visits. The recruitment strategy will be deemed 'feasible' if 15 participants are recruited within the 8 weeks.
Time Frame: Baseline; Week 8
Population: 60 participants were screened for eligibility. 43 were excluded (12 did not meet eligibility criteria; 31 declined to participate). 17 consented and 16 completed initial baseline visits. 13 decided to participate in the intervention. 11 received the allocated intervention and 2 did not (dropped out due to time constraints). Demographic variables were assessed among intervention participants, explaining the discrepancies between the results and participant flow sections.
Measure: Count of Participants; unit: Participants
Arm/Group | ABT Weight Loss Intervention
Number analyzed (Participants) | 60
Participants | 16

2. Primary Outcome: Percentage of Participants Who Did Not Complete the Intervention.
Description: The attrition strategy will be deemed "feasible" if there is less than 50% attrition at the end of the 6-month intervention. This percentage details attrition, or the percentage of participants who did not complete the intervention.
Time Frame: Baseline; Month 6
Population: 17 participants consented; 16 participants completed the 2 initial baseline clinic visits. Of the 16 participants who completed baseline visits, 13 decided to participate in the intervention. 11 received the allocated intervention and 2 did not (dropped out due to time constraints). Demographic variables were assessed among intervention participants (n=13).This explanation provides insights to the discrepancies between the results and participant flow sections.
Measure: Number; unit: percentage of participants
Arm/Group | ABT Weight Loss Intervention
Number analyzed (Participants) | 13
percentage of participants | 15.4

3. Primary Outcome: Percentage of Participants Who Decide to Participate in the Intervention
Description: Of the participants who completed baseline visits, this percentage details what percentage of enrollees decided to participate in the intervention. The study will be deemed "acceptable" if at least 80% of enrolled participants decide to participate in the intervention.
Time Frame: Baseline; Week 1
Population: 17 participants consented; 16 participants completed the 2 initial baseline visits. Of the 16 participants who completed baseline visits, 13 decided to participate in the intervention. Of the 13 participants who decided to participate in the intervention, 11 received the allocated intervention and 2 dropped out due to time constraints. This explanation provides insight to discrepancies between the results and participant flow.
Measure: Number; unit: percentage of participants
Arm/Group | ABT Weight Loss Intervention
Number analyzed (Participants) | 16
percentage of participants | 81.3

4. Primary Outcome: Percentage of Participants Who Attend All Intervention Sessions.
Description: This percentage details the percentage of those who attended all 15 intervention sessions among intervention completers (n=11). The study will be deemed 'acceptable' if at least 70% of intervention completers attend all sessions.
Time Frame: Week 1; Week 24
Population: 17 participants consented; 16 participants completed the 2 initial baseline clinic visits. Of the 16 participants who completed baseline visits, 13 decided to participate in the intervention. Of the 13 participants who decided to participate in the intervention, 11 received the allocated intervention and 2 did not (dropped out due to time constraints). This explanation provides insight into discrepancies between the results
Measure: Number; unit: percentage of participants
Arm/Group | ABT Weight Loss Intervention
Number analyzed (Participants) | 11
percentage of participants | 90.9

5. Secondary Outcome: Change in BMI Z-score
Description: Body mass index (BMI) z-scores are measures of weight adjusted for the height, age, and sex of the child. BMI z-scores correspond with growth chart percentiles. These scores are calculated with an external reference rather than internal references. In this study, the Centers for Disease Control and Prevention SAS program was used to calculate scores based on 2000 CDC growth charts. Additionally, a clinically significant change in BMI z-score was defined as greater than or equal to -0.15 as this decrease has shown improvements in one or more cardiovascular disease risk factor. The central z-score value is 0, representing the population mean, and standard deviations below the mean indicate better outcomes.
Time Frame: Baseline; Month 6
Population: 17 participants consented; 16 participants completed the 2 initial baseline clinic visits. Of the 16 participants who completed baseline visits, 13 decided to participate in the intervention. Of the 13 participants who decided to participate in the intervention, 11 received the allocated intervention and 2 did not (dropped out due to time constraints). This explanation provides insight into any discrepancies between the participant flow and results sections.
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | ABT Weight Loss Intervention
Number analyzed (Participants) | 11
z-scores | -0.15 (0.34)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of baseline through study completion [6 months].
Arm/Group | ABT Weight Loss Intervention
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03284788/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03284788/ICF_001.pdf